CLINICAL TRIAL: NCT06371222
Title: Role of Ivabradine on Heart Rate and Quality of Life in Patients With Mitral Stenosis in Sinus Rhythm - a Randomized Control Trial
Brief Title: Role of Ivabradine on Heart Rate and Quality of Life in Patients With Mitral Stenosis in Sinus Rhythm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Skeikh Foyez Ahmed, consultant cardilogist, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BSMMU/2023/6502
Record Dates: First submitted 2024-03-19; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Mitral Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis | interventions — Ivabradine; Adrenergic beta-Antagonists; Metoprolol

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled group (Active Comparator): controlled group
  Interventions: Drug: Beta blocker
- intervention group (Experimental): intervention group
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — 5 mg for 3 months
  Arms: intervention group
Drug: Beta blocker — controlled group
  Other Names: metoprolol
  Arms: controlled group

SUMMARY:
Mitral stenosis, a condition characterized by narrowing of the mitral valve orifice, remains a significant cause of morbidity and mortality worldwide, particularly in regions where rheumatic fever is endemic. Despite advancements in medical and surgical management, patients with mitral stenosis often suffer from symptoms such as dyspnea, fatigue, and reduced exercise tolerance, significantly impacting their quality of life (QoL) [1].

One of the hallmark features of mitral stenosis is the development of sinus rhythm, which can be associated with elevated heart rates due to decreased diastolic filling time and compensatory mechanisms to maintain cardiac output. Persistent tachycardia in patients with mitral stenosis contributes to increased myocardial oxygen demand, exacerbating symptoms and potentially leading to adverse outcomes [2].

In recent years, ivabradine, a selective inhibitor of the If current in the sinoatrial node, has emerged as a promising therapeutic option for controlling heart rate in various cardiovascular conditions, including chronic heart failure and ischemic heart disease [3]. By specifically targeting the cardiac pacemaker cells, ivabradine reduces heart rate without affecting myocardial contractility or conduction, offering a unique mechanism of heart rate control compared to traditional beta-blockers or calcium channel blockers [4].

However, the role of ivabradine in patients with mitral stenosis in sinus rhythm remains uncertain, and there is limited evidence regarding its efficacy and impact on QoL in this specific patient population. Therefore, the aim of this randomized controlled trial (RCT) is to investigate the effects of ivabradine on heart rate control and QoL in patients with mitral stenosis in sinus rhythm.

DETAILED DESCRIPTION:
Symptoms of mitral stenosis (MS) are may be sometimes cause significant risk mainly during increase heart and exercise. Beta-blockers are given in some patients for heart rate (HR) in MS, which in turn improve the symptoms, but they have side effects. Ivabradine has a selective action on the sinus node with less side effects. Some studies have recently investigated the role of ivabradine in MS in sinus rhythm. We will determine the efficacy and safety status of ivabradine, compared to standard treatment on maximum HR achieved among patients in sinus rhythm with MS as well as the impact of drug treatment on QOL.

Research question:

What is the role of ivabradine in comparison with standard treatment (beta blocker) on heart rate in sinus rhythm and quality of life in mitral stenosis patients?

Aims and Objectives:

General:

To assess and compare the status of ivabradine with beta blocker on heart rate in sinus rhythm in mitral stenosis patients

Specific:

1. To evaluate the effect of ivabradine on heart rate at base line and after 3 months in sinus rhythm mitral stenosis patients
2. To assess the comparative efficacy of ivabradine versus beta blocker on heart rate at baseline and after 3 months in sinus rhythm in mitral stenosis patients
3. To assess the comparative safety of ivabradine and beta blocker in sinus rhythm in mitral stenosis patients
4. To assess & compare the effect of ivabradine with beta blocker on quality of life in sinus rhythm mitral stenosis patients

Additional Objective

• To measure LVEF by bedside 2D & M mode echocardiography

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* sex- male and females
* MS patients admitted to BSMMU
* All patients who will give written informed consent
* Diagnosis of Mitral stenosis by ECG & Echo
* Mitral stenosis patients with heart rate above 80bpm
* trans thoracic echocardiography mitral valve area >1.5 cm2

Exclusion Criteria:

* Significant others valvular or congenital heart disease
* Prior history of MI, Coronary intervention or CABG
* Heart failure
* Previous cardiac surgery
* Any form of cardiomyopathy
* Conduction defect
* Haemodynamically unstable patient and patient with an unstable co-morbid illness
* Renal impairment
* COVID-19 patient
* Urgent need for surgical treatment or balloon valvoplasty
* Patients who have indication for surgical treatment or BMV
* Heart failure
* Sick sinus syndrome patients
* Pregnancy
* Atrial fibrillation
* Patient with blood pressure systolic < 90 and diastolic < 50 mm of Hg

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
effect of ivabradine in MS patients | three months
  effect of ivabradine from baseline with the study drugs on heart rate

SECONDARY OUTCOMES:
quality of life of MS patients | three months
  Questionnaire to assess quality of life changes

CONTACTS AND LOCATIONS:
Overall Officials: sheikh dr ahmed, MD, Principal Investigator — BSMMU, DHAKA
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No